CLINICAL TRIAL: NCT02706704
Title: Efficacy of Intravitreal Adalimumab Compared to Subcutaneous Adalimumab in Patients With Non-infectious Uveitis
Brief Title: Intravitreal Adalimumab Versus Subcutaneous Adalimumab in Non-infectious Uveitis
Acronym: IVAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPH.RH.07
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Uveitis; Non-Infectious Uveitis
Keywords: Intravitreal Adalimumab; Subcutaneous Adalimumab
MeSH Terms: conditions — Uveitis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravitreal (Active Comparator): Intravitreal injection of 1.5mg/0.03ml adalimumab given at zero, 2 weeks, and then every 4 weeks.
  Interventions: Drug: Adalimumab
- Systemic (Active Comparator): Subcutaneous injection of 40 mg adalimumab (Humira) given every 2 weeks.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
The objective of this study is to compare and evaluate the efficacy of subcutaneous (40mg) adalimumab biweekly injections to intravitreal adalimumab (1.5 mg/ 0.03 mL) administration, given at zero, 2 weeks then every four weeks, in subjects with active non-infectious intermediate-, posterior-, or pan-uveitis.

DETAILED DESCRIPTION:
Subject groups:

32 subjects will be enrolled in this study, 16 in each arm. They will be randomized to receive either 1.5 mg/ 0.03 mL of adalimumab by intravitreal injection or 40 mg of adalimumab subcutaneously at their first treatment visit and at the 2 weeks visit if eligible for a repeat injection. Follow up will be every 2 days the first week then one week later and after that every 4-week intervals for total of 26 weeks.

Intervention Details:

* Systemic adalimumab: Subcutaneous injection of 40 mg adalimumab (Humira) given every 2 weeks.
* Local adalimumab: Intravitreal injection of 1.5mg/0.03ml adalimumab given at zero, 2 weeks, and then every 4 weeks.

Pre-treatment work up

Patients will undergo a comprehensive eye exam:

* Visual acuity, slit-lamp examination of the anterior segment, dilated fundus examination, electroretinography (ERG) and fluorescein angiography (FA).
* Central macular thickness of all eyes will be measured with ocular coherence tomography before treatment.
* Purified Protein Derivative (PPD), Complete blood count (CBC) and SGPT.

Post-injection follow-up

* Patients will be followed up every 2 days during the first week then one week later and after that every 4-week intervals.
* On follow up visits, if deterioration in vision of two or more ETDRS lines or worsening of ocular inflammation by more than 1+ cells/haze is detected at any visit, patients will be removed from the study and receive appropriate treatment. Otherwise, if vision was stable or improved and/or inflammation is same or better, patients will be re-injected.
* Follow up is for 26 weeks.
* OCT and fluorescein angiography each visit.
* ERG will be performed at baseline and 26 weeks.
* Blood studies (CBC and SGPT) will be performed at baseline, 14 weeks and at 26 weeks.
* Injections would be delayed if a patient has an acute infection and would be given when it subsides.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age.
* Subject is diagnosed with non-infectious intermediate-, posterior-, or pan-uveitis.
* Subject must have active disease at baseline as defined by the presence of at least 1 of the following parameters in at least one eye despite at least 2 weeks of prednisone ≥ 10 mg/day (or oral corticosteroid equivalent):

  * Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion
  * ≥ 1+ anterior chamber cells (Standardization of Uveitis Nomenclature [SUN] criteria)
  * ≥ 1+ vitreous haze (National Eye Institute [NEI]/SUN criteria)
* Subject with documented prior adequate response to oral corticosteroids (equivalent of oral prednisone up to 1 mg/kg/day).
* If subject is on prednisone >=10 mg (or corticosteroid equivalent) at baseline, the dose has not been increased or decreased in the past 14 days.
* No increase in the immune modulatory therapy in the past three months
* Negative PPD test.
* Positive PPD test on anti Tb medications.

Exclusion Criteria:

* Subject with isolated anterior uveitis.
* Subject with confirmed or suspected infectious uveitis, including but not limited to infectious uveitis due to TB, cytomegalovirus, lyme disease, toxoplasmosis and herpes simplex virus (HSV).
* Subject with serpiginous choroidopathy.
* Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial.
* Subject with corneal or lens opacities that preclude the evaluation of the vitreous haze.
* Subject with uncontrolled high intraocular pressure of ≥ 25 mmHg on maximal therapy.
* Subject with intermediate uveitis and symptoms and/or MRI findings suggestive of a demyelinating disease such as multiple sclerosis. All subjects with intermediate uveitis must have had a prior brain MRI at time of or after diagnosis of intermediate uveitis.
* Subject has received glucocorticosteroids implant (Retisert®), or Ozurdex within 6 months prior to baseline visit.
* Subject has received intraocular or periocular corticosteroids or intravitreal methotrexate within 90 days prior to Baseline visit.
* Subject with proliferative or severe non-proliferative diabetic retinopathy.
* Subject with neovascular/wet age-related macular degeneration
* Subject with abnormality of vitreo-retinal interface (i.e., vitreomacular traction, epiretinal membranes, etc.) with the potential for macular structural damage independent of the inflammatory process.
* Subject with a systemic inflammatory disease and requires additional therapy with a systemic immunosuppressive agent at the time of study entry.
* Subjects with history of active or latent Mycobacterium tuberculosis documented by Purified Protein Derivative (PPD) and chest X-ray and not anti tuberculosis (TB) treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Vitreous Haze | 26 Weeks
  Change in Vitreous Haze grade in each eye [National Eye Institute (NEI)/ Standardization of Uveitis Nomenclature (SUN) criteria]
Anterior Chamber Cells | 26 Weeks
  Change in Anterior Chamber (AC) cell grade in each eye.

SECONDARY OUTCOMES:
Visual Acuity | 26 Weeks
  Change in ETDRS letters and logarithm of the minimum angle of resolution (log MAR) best-corrected visual acuity (BCVA) in each eye.
Macular Edema | 26 Weeks
  Change in central retinal thickness on Optical Coherence Tomography (OCT).
Angiography Score | 26 Weeks
  Change in fluorescein angiography score
Steroids Tapering | 26 Weeks
  If the patient is initially on steroids (pre-enrolment); Success in tapering steroid dose as a response to the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Rola N Hamam, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamam RN, Barikian AW, Antonios RS, Abdulaal MR, Alameddine RM, El Mollayess G, Mansour AM. Intravitreal Adalimumab in Active Noninfectious Uveitis: A Pilot Study. Ocul Immunol Inflamm. 2016 Jun;24(3):319-26. doi: 10.3109/09273948.2014.990041. Epub 2014 Dec 30. PMID 25549063
- [Background] Santos Lacomba M, Marcos Martin C, Gallardo Galera JM, Gomez Vidal MA, Collantes Estevez E, Ramirez Chamond R, Omar M. Aqueous humor and serum tumor necrosis factor-alpha in clinical uveitis. Ophthalmic Res. 2001 Sep-Oct;33(5):251-5. doi: 10.1159/000055677. PMID 11586057
- [Background] Perez-Guijo V, Santos-Lacomba M, Sanchez-Hernandez M, Castro-Villegas Mdel C, Gallardo-Galera JM, Collantes-Estevez E. Tumour necrosis factor-alpha levels in aqueous humour and serum from patients with uveitis: the involvement of HLA-B27. Curr Med Res Opin. 2004;20(2):155-7. doi: 10.1185/030079903125002847. PMID 15006008
- [Background] Rudwaleit M, Rodevand E, Holck P, Vanhoof J, Kron M, Kary S, Kupper H. Adalimumab effectively reduces the rate of anterior uveitis flares in patients with active ankylosing spondylitis: results of a prospective open-label study. Ann Rheum Dis. 2009 May;68(5):696-701. doi: 10.1136/ard.2008.092585. Epub 2008 Jul 28. PMID 18662932
- [Background] Mansour AM. Adalimumab in the therapy of uveitis in childhood. Br J Ophthalmol. 2007 Mar;91(3):274-6. doi: 10.1136/bjo.2006.108050. PMID 17322463
- [Background] Diaz-Llopis M, Garcia-Delpech S, Salom D, Udaondo P, Hernandez-Garfella M, Bosch-Morell F, Quijada A, Romero FJ. Adalimumab therapy for refractory uveitis: a pilot study. J Ocul Pharmacol Ther. 2008 Jun;24(3):351-61. doi: 10.1089/jop.2007.0104. PMID 18476805
- [Background] Wu L, Hernandez-Bogantes E, Roca JA, Arevalo JF, Barraza K, Lasave AF. intravitreal tumor necrosis factor inhibitors in the treatment of refractory diabetic macular edema: a pilot study from the Pan-American Collaborative Retina Study Group. Retina. 2011 Feb;31(2):298-303. doi: 10.1097/IAE.0b013e3181eac7a6. PMID 21099452
- [Background] Androudi S, Tsironi E, Kalogeropoulos C, Theodoridou A, Brazitikos P. Intravitreal adalimumab for refractory uveitis-related macular edema. Ophthalmology. 2010 Aug;117(8):1612-6. doi: 10.1016/j.ophtha.2009.12.011. Epub 2010 Apr 8. PMID 20378179
- [Background] Manzano RP, Peyman GA, Carvounis PE, Damico FM, Aguiar RG, Ioshimoto GL, Ventura DF, Cursino ST, Takahashi W. Toxicity of high-dose intravitreal adalimumab (Humira) in the rabbit. J Ocul Pharmacol Ther. 2011 Aug;27(4):327-31. doi: 10.1089/jop.2010.0174. Epub 2011 Jun 13. PMID 21668348
- [Background] Tsilimbaris M, Diakonis VF, Naoumidi I, Charisis S, Kritikos I, Chatzithanasis G, Papadaki T, Plainis S. Evaluation of potential retinal toxicity of adalimumab (Humira). Graefes Arch Clin Exp Ophthalmol. 2009 Aug;247(8):1119-25. doi: 10.1007/s00417-009-1065-y. Epub 2009 Mar 19. PMID 19296122
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117